CLINICAL TRIAL: NCT03224897
Title: Effects of Transcranial Direct Current Stimulation Over the Left Ventrolateral Prefrontal Cortex on Cognitive Reappraisal
Brief Title: Effects of Transcranial Direct Current Stimulation Over the Left VLPFC on Cognitive Reappraisal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Effects of Transcranial Direct Current Stimulation Over the Left Ventrolateral Prefrontal Cortex on Cognitive Reappraisal, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: tDCS_VLPFC_Reappraisal
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Reappraisal; Emotion Regulation; tDCS; Reinterpretation
MeSH Terms: conditions — Emotional Regulation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The 60 participants will be divided into 3 groups: anodal, cathodal and sham stimulation. While receiving the transcranial direct current (tDCS) stimulation, participants will perform a reappraisal task. Four series of 15 IAPS pictures will be randomly passed on a computer screen. 3 of the 4 sets of pictures contain negative pictures, matched according to valence and arousal of the IAPS norm ratings (p<0.05) and were assigned to one of instruction condition (upregulate, downregulate or maintain). The other set will contain neutral pictures with the instruction maintain. Participants will be asked to apply the instruction assigned to each picture and then rank the intensity of negative emotional arousal felt after using the reappraisal strategy, varying from 1 (weak) to 7 (strong). ANOVA will be used to compare the median subjective emotion intensity evaluation for each strategy intra-subjects and inter-groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The tDCS device was placed at the back of the participants, so they could not see the parameters of stimulation. The participants of the sham stimulation group received anode stimulation for 30s, and then the device was turned off. The participants feel the initial itching in all conditions, so the are not able to distinguish to which condition of stimulation they are submitted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cathodal tDCS (Active Comparator)
  Interventions: Device: Cathodal tDCS
- Anodal tDCS (Active Comparator)
  Interventions: Device: Anodal tDCS
- Sham tDCS (Sham Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Cathodal tDCS — Volunteers will be submitted to 1,0 mA cathodal stimulation during experiment. The stimulation will be applied through a pair of saline-soaked surface sponge electrodes for 20 minutes, with a 10s ramp up and down. The 4,5 x 5,0 cm "active" electrode will be placed over the crossing point between Fz-T3 and F7-Cz and the 12 x 5 cm "return" electrode will be placed over Fp2 according to the 10-20 EEG system.
  Arms: Cathodal tDCS
Device: Anodal tDCS — 1,0mA anodal stimulation will be applied through a pair of saline-soaked surface sponge electrodes for 20 minutes, with a 10s ramp up and down. The 4,5 x 5,0 cm "active" electrode will be placed over the crossing point between Fz-T3 and F7-Cz and the 12 x 5 cm "return" electrode will be placed over Fp2 according to the 10-20 EEG system.
  Arms: Anodal tDCS
Device: Sham tDCS — 1,0 mA anodal stimulation will be applied through a pair of saline-soaked surface sponge electrodes for 30 seconds, with a 10s ramp up and down. The 4,5 x 5,0 cm "active" electrode will be placed over the crossing point between Fz-T3 and F7-Cz and the 12 x 5 cm "return" electrode will be placed over Fp2 according to the 10-20 EEG system. The participant will not know when the stimulator is turned off and will continue to perform the experimental task as in the other groups.
  Arms: Sham tDCS

SUMMARY:
This study aims to investigate the role of the left ventrolateral prefrontal cortex (VLPFC) on cognitive reappraisal, using the reinterpretation strategy. For this purpose, we will produce direct disturbance to the activity of this area through anodal and cathodal transcranial direct current stimulation during a reinterpretation task.

A double-blind randomized sham-controlled trial will be conducted. 60 healthy volunteers will be allocated into three groups. Each group will receive one type of stimulation (anodal, cathodal or sham) while accomplishing a cognitive task on reinterpretation using images from the International Affective Pictures System (IAPS). The task consists in applying a given emotional regulation condition (downregulate, upregulate or maintain emotions) to a series of images and ranking the intensity of the emotional arousal felt after doing this procedure to each picture. The effects of tDCS on the subjective evaluation of emotional arousal after reinterpretation in each group will be compared.

DETAILED DESCRIPTION:
60 healthy graduation and post-graduation at the Federal University of Pernambuco (UFPE) students will take part of the study. After providing written informed consent, the volunteers will respond to four online questionnaires, received by email: a sociodemographic questionnaire investigating eligibility conditions; the brazilian version of the Self-Reporting Questionnaire (SRQ-20) to screen for common psychiatric disorders; the brazilian self-report version of the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) 3.0, to screen for drug-related disorders; and the brazilian version of the Emotion Regulation Questionnaire (ERQ) to evaluate individual profile of habitual use of emotion regulation strategies. They will be oriented to contact to researchers if they have any doubts. After filling the questionnaires, the volunteers will be contacted to be informed about eligibility. Individuals with previous history of epilepsy/ convulsions, brain tumors, neurosurgery, or with brain metallic implants or pacemakers, as well as in current use of psychotropic medication will be excluded from the study. The volunteers that score less than 5 point in SRQ-20 or more than 10 points for alcohol or more than 3 points for other substances in self-report ASSIST 3.0 will also be excluded from the sample.

The selected volunteers will receive a training on the cognitive task. Firstly, they will receive a brief explanation and examples on cognitive reappraisal, the reinterpretation strategies and the instructions. Against the instruction MAINTAIN, they should simply look at the pictures and maintain their emotional experience, according to their initial interpretation of the presented situation. When facing the instruction DOWNREGULATE, they should look to the picture and imagine that the situation is better or will become better than initially perceived and when instructed to UPREGULATE, they should look to the picture and imagine that the situation is worse or will become worse than initially perceived. They will be presented on the computer screen to a series of 21 negative images preceded of a screen containing one of instructions (7 images for each instruction) and 7 neutral images preceded of a screen with the instruction maintain. The images will be presented randomly and they will be asked to generate strategies to each situation. They will be guided to provide adequate strategies to the received instructions and will receive a standardized example for each picture. After this phase, they will be presented to the same series of images in the same format as the experimental cognitive task. They will see 4 screens for each picture, following uninterruptedly. The fist will contain the strategy for 2 seconds, the second will present the picture for 8 seconds, the third will contain a visual scale from 1-7 to rank the intensity of the emotional arousal felt after applying the strategy to the picture (1=very weak; 7=very strong). They will be asked to press the correspondent number on a numerical keyboard into 5 seconds. The final screen will have the instruction RELAX for 3 seconds and they should wait and relax until the subsequent task initiate.

The experiment will be conducted 3-5 days later. Before the experiment, the participant will respond to 2 questionnaires: the first will investigate behaviors that could influence the results of the experiment (sleep, psychostimulant substance intake) and the second will evaluate the current momentaneous status of the volunteer (humor, attention, fatigue). After a brief training of the cognitive task with 6 pictures, we will proceed to the electrodes montage. tDCS (1 mA) will be applied through a pair of saline-soaked surface sponge electrodes connected to a battery-driven constant current stimulator and positioned according to the 10-20 EEG system over the left VLPFC. A 4,5x4cm "active" electrode will be placed over the crossing point between T3-Fz and F7- Cz and a 12x5cm "return" electrode will be positioned over Fp2. The big return electrode will be used to attenuate the effects of stimulation over that region. The stimulation will start 4 minutes before the beginning of the cognitive task. The participants of the real stimulation groups will receive stimulation for 20 minutes, with 10 seconds ramp-up and down periods. In the sham group, the participants will receive the stimulation for 30 seconds.

Measures of central tendency and dispersion (mean and standard deviation) for continuous variables and measures of frequency for the categorical variables will be used in the sample characterization. T-test for independent samples or qui-square will be used to verify comparability between groups for continuous and categorical variables, respectively. Shapiro-Wilk test will be used to evaluate normality. Repeated measures analyses of variance (ANOVAs) will be used to test for main effects and interaction with the within subjects factors regulation condition (downregulate, upregulate, negative maintain, neutral maintain) and the between-subjects factors (anodal, cathodal, sham stimulation) in case of normality. Paired t-test will be used for compare intra-group differences. T-test for independent samples will be conducted to compare inter-group differences. The sphericity will be verified with the Mauchly's test. Greenhouse-Geisser correction will be used when necessary. If normality is not verified, Friedman's test with post-hoc Wilcoxon test will be conducted to detect intra-group differences and post-hoc Mann-Whitney test will be conducted for inter-group differences. Two-tailed tests will be performed at 95% confidence interval for all analyses. Statistical analyses will be carried out using SPSS (Statistical Package for Social Sciences) 20.0 version for Windows (SPSS Inc, Chicago IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* graduate and post-graduate students at UFPE
* aged > 18 years-old

Exclusion Criteria:

* seizures antecedent
* brain tumor
* neurosurgery antecedent
* metalic implant on the head
* cardiac pacemaker
* current psychotropic usage
* SRQ-20 score > 5
* ASSIST 3.0 (sum from 2-7 questions) > 10 for alcohol or > 3 for other drugs
* left-handed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Subjective Emotional Arousal Rating | 20 minutes
  The rating from 1-7 (1=very weak; 7=very strong) of the negative emotional arousal felt by the volunteer after the volunteer after using the reappraisal strategy for each picture.

SECONDARY OUTCOMES:
Self-evaluation about the success in performing cognitive task | 20 minutes
  Self-evaluation of success in performing adequately the cognitive task in a 1-9 likert scale (0=no success; 9=total success)

OTHER OUTCOMES:
ERQ Questionnaire score | 20 minutes
  The scores for the use of both strategies - reappraisal and suppression in the ERQ questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Applied Neuroscience Laboratory, Recife, Pernambuco
  - Federal University of Pernambucano, Recife, Pernambuco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feeser M, Prehn K, Kazzer P, Mungee A, Bajbouj M. Transcranial direct current stimulation enhances cognitive control during emotion regulation. Brain Stimul. 2014 Jan-Feb;7(1):105-12. doi: 10.1016/j.brs.2013.08.006. Epub 2013 Sep 21. PMID 24095257
- [Background] Ochsner KN, Ray RD, Cooper JC, Robertson ER, Chopra S, Gabrieli JD, Gross JJ. For better or for worse: neural systems supporting the cognitive down- and up-regulation of negative emotion. Neuroimage. 2004 Oct;23(2):483-99. doi: 10.1016/j.neuroimage.2004.06.030. PMID 15488398
- [Background] Cattaneo Z, Pisoni A, Papagno C. Transcranial direct current stimulation over Broca's region improves phonemic and semantic fluency in healthy individuals. Neuroscience. 2011 Jun 2;183:64-70. doi: 10.1016/j.neuroscience.2011.03.058. Epub 2011 Apr 6. PMID 21477637
- [Background] Pisoni A, Papagno C, Cattaneo Z. Neural correlates of the semantic interference effect: new evidence from transcranial direct current stimulation. Neuroscience. 2012 Oct 25;223:56-67. doi: 10.1016/j.neuroscience.2012.07.046. Epub 2012 Jul 31. PMID 22863670
- [Background] Cohen-Maximov T, Avirame K, Floel A, Lavidor M. Modulation of Gestural-verbal Semantic Integration by tDCS. Brain Stimul. 2015 May-Jun;8(3):493-8. doi: 10.1016/j.brs.2014.12.001. Epub 2014 Dec 11. PMID 25558040